CLINICAL TRIAL: NCT05917977
Title: A Randomized Controlled Study of Collective Motivational Interviewing (CMI) for Adolescents With Internet Gaming Disorder
Brief Title: Collective Motivational Interviewing (CMI) for Adolescents With Internet Gaming Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong College of Technology (Other)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other); Nottingham Trent University (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Dr. Tse Ka Wo, BSW HKU, MSc International Addiction Studies KCL, Ph.D. HKU, MINT Certified Trainer, CGC (Canada), Ccoun&AF(HKPCA), R.S.W. (Hong Kong), Assistant Professor, Department of Applied Social Sciences, Hong Kong College of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGC/FDS21/H01/22
Record Dates: First submitted 2023-05-09; First posted 2023-06-26 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Internet Gaming Disorder
Keywords: Motivational interviewing; Family counselling; Effective treatment; Randomized controlled trial
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The present study adopted a two-armed RCT to examine the efficacy of CMI in improving IGD among adolescents with IGD. The research participants will be randomly assigned to either the intervention group (four-session CMI intervention plus IGD educational materials) or the control group (IGD education materials alone). Block randomization will be executed, of which the block size is 4. Computer-generated randomization allocation codes will be produced and sealed in opaque envelopes by a research associate with no involvement in recruitment. One envelope will be drawn and opened by the project officer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Education Materials) (Other): After completing the baseline screening, survey and randomization, the participants in the control group will receive educational materials regarding topics including: (1) what IGD is and its consequences, (2) how to communicate with parents about the gaming time, and (3) how to develop a healthy lifestyle, etc.
  Interventions: Other: Control group (Education Materials)
- Intervention group (Collective Motivational Interviewing plus Education Materials) (Experimental): Participants in the intervention group will be given the same Internet Gaming Disorder (IGD) education materials as those in the control group, thus, they will further participate in four counseling sessions with Collective Motivational Interviewing (CMI) (each session 60 mins). In the first session, adolescents with Internet Gaming Disorder will be implemented a standard MI session to elicit and strengthen the client's motivation to change. In the second session, a nominated CSO of the client will participate in a standard MI session to elicit their motivation to help the client toward change and prepare positive attitudes of CSO for the conjoint session. Afterward, the third and fourth sessions (75 mins) will be conjoint sessions. The Collective Motivational Interviewing practitioners will create a safe platform for both parties to share their perspectives with openness and trustfulness, in turn, to reach an agreed goal (e.g., develop a change plan on internet gaming behaviors).
  Interventions: Behavioral: Collective Motivational Interviewing plus Education Materials

INTERVENTIONS:
Behavioral: Collective Motivational Interviewing plus Education Materials — The participants in the intervention group will receive IGD educational materials as well as four counseling sessions of CMI intervention.
  Arms: Intervention group (Collective Motivational Interviewing plus Education Materials)
Other: Control group (Education Materials) — The participants in the control group will receive IGD educational materials.
  Arms: Control group (Education Materials)

SUMMARY:
The present study examines the efficacy of CMI in reducing adolescent IGD symptoms and enhancing social support given by CSOs among adolescents with high risk of IGD (probable IGD cases screened positive by validated tools). It is hypothesized that the intervention group (with CMI plus IGD education materials for both the clients and his/her selected CSO) would show more improvements in reduction in the severity of IGD, motivation to change maladaptive gaming behaviour, craving on gaming, and social support obtained from CSOs than to the control group (only educational materials for both the client and the CSOs).

DETAILED DESCRIPTION:
This study adopts a randomized controlled efficacy study with an open-label parallel-group design. The trial will be registered by the WHO's International Clinical Trials Registry Platform once the project is approved. Research participants will be recruited from the primary and secondary schools, and youth social services. After completing the screening process, research participants who are confirmed to fit the inclusion criteria will be randomly assigned to the intervention group with CMI intervention plus IGD education materials to both adolescents with IGD and their CSO or the control group with IGD education materials alone. The present study sets four-time points to track the change in the between-group difference of the primary and secondary outcomes from the baseline (T0) to post-intervention (T1), 3-month follow-up (T2), and 6-month follow-up (T3).

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* Aged between 10-16
* Probable IGD condition screened by the Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) reaching the cut-off value at 21, those at high risk of having IGD but no IGD cases with clinical diagnosis, although the symptoms measured by IGDS9-SF are equivalent to DSM-5 IGD criteria)
* Hong Kong ID card holder
* Chinese speaking
* Student identity
* Possessing an electronic mobile device or computer
* Willingness to participate in the intervention/control group and complete four surveys (baseline, post-intervention, 3-month follow-up, and 6-month follow-up)
* Can nominate a CSO (e.g., parents) [client's autonomy is a critical factor to facilitate motivation posited by the self-determination theory (Ryan & Deci, 2020) (9) to obtain informed consent and parental consent

Inclusion Criteria for CSO:

* Aged greater than 18 years
* Having a close relationship with the adolescent with probable IGD (as rated by participants being generally supportive of the participants)
* Being willing to participate in the present study and provide informed consent

Exclusion Criteria for Adolescents:

* Participants who have psychiatric problems such as psychosis, significant cognitive impairment and/or receiving active and structured psychotherapy about IGD elsewhere will be excluded (Nielsen et al., 2021).

Exclusion Criteria for CSO:

* Participants who have psychosis, aggressive or suicidal behavior
* Having life-threatening medical conditions

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of IGD | Change from Baseline (T0) Severity of IGD at posttest (T1: After intervention)
  The nine-item Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) are used to detect the change in the severity of IGD. It is the first brief standardized psychometric tool of IGD based on the nine DSM-5 IGD criteria. This instrument has been translated into 15 languages and is widely used in research and clinical settings. In addition, a validated Chinese version with satisfactory psychometric properties is available (Qin et al., 2020). The items were rated by using a 5-point Likert scale (1 = Never to 5 = Very often).
Severity of IGD | Change from Baseline (T0) Severity of IGD at 3-month follow-up (T2)
  The nine-item Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) are used to detect the change in the severity of IGD. It is the first brief standardized psychometric tool of IGD based on the nine DSM-5 IGD criteria. This instrument has been translated into 15 languages and is widely used in research and clinical settings. In addition, a validated Chinese version with satisfactory psychometric properties is available (Qin et al., 2020). The items were rated by using a 5-point Likert scale (1 = Never to 5 = Very often).
Severity of IGD | Change from Baseline (T0) Severity of IGD at 6-month follow-up (T3)
  The nine-item Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) are used to detect the change in the severity of IGD. It is the first brief standardized psychometric tool of IGD based on the nine DSM-5 IGD criteria. This instrument has been translated into 15 languages and is widely used in research and clinical settings. In addition, a validated Chinese version with satisfactory psychometric properties is available (Qin et al., 2020). The items were rated by using a 5-point Likert scale (1 = Never to 5 = Very often).

SECONDARY OUTCOMES:
Motivation to change maladaptive gaming behaviour | Change from Baseline (T0) Motivation to change maladaptive gaming behaviour at posttest (T1: After intervention)
  Contemplation Ladder for Internet Gaming (CL-LG), which is derived from the Contemplation Ladder measure the motivation to quit smoking (Biener & Abrams, 1991), are employed. Contemplation Ladder for drug use problems is commonly used in clinical settings and research in Hong Kong (Siu et al., 2018). The instrument measures the motivation to abstain from maladaptive gaming behaviors based on a single brief option of 11 rungs and five types of statements. The instrument is rated on a scale from 0 to 10, with each point representing a specific statement showing a corresponding stage of change. The ladder has been used in smoking cessation studies, which displayed strong reliability and validity with strong intercorrelations (Pearson's r = .82 - .98) (Rustin & Tate, 1993).
Motivation to change maladaptive gaming behaviour | Change from Baseline (T0) Motivation to change maladaptive gaming behaviour at 3-month follow-up (T2)
  Contemplation Ladder for Internet Gaming (CL-LG), which is derived from the Contemplation Ladder measure the motivation to quit smoking (Biener & Abrams, 1991), are employed. Contemplation Ladder for drug use problems is commonly used in clinical settings and research in Hong Kong (Siu et al., 2018). The instrument measures the motivation to abstain from maladaptive gaming behaviors based on a single brief option of 11 rungs and five types of statements. The instrument is rated on a scale from 0 to 10, with each point representing a specific statement showing a corresponding stage of change. The ladder has been used in smoking cessation studies, which displayed strong reliability and validity with strong intercorrelations (Pearson's r = .82 - .98) (Rustin & Tate, 1993).
Motivation to change maladaptive gaming behaviour | Change from Baseline (T0) Motivation to change maladaptive gaming behaviour at 6-month follow-up (T3)
  Contemplation Ladder for Internet Gaming (CL-LG), which is derived from the Contemplation Ladder measure the motivation to quit smoking (Biener & Abrams, 1991), are employed. Contemplation Ladder for drug use problems is commonly used in clinical settings and research in Hong Kong (Siu et al., 2018). The instrument measures the motivation to abstain from maladaptive gaming behaviors based on a single brief option of 11 rungs and five types of statements. The instrument is rated on a scale from 0 to 10, with each point representing a specific statement showing a corresponding stage of change. The ladder has been used in smoking cessation studies, which displayed strong reliability and validity with strong intercorrelations (Pearson's r = .82 - .98) (Rustin & Tate, 1993).
Craving for Internet Gaming | Change from Baseline (T0) Craving for Internet Gaming at posttest (T1: After intervention)
  Craving for Internet Gaming Scale (CIGS) is used to measure respondents' intensity, frequency, duration of their craving, and capability to resist acting on their craving for a particular period of time. It comprises five-item, scoring from 0 to 6 for each item. Respondents with higher scores tend to have higher levels of gaming craving (Cronbach's alpha was .88-.91) (Savci & Griffiths, 2019).
Craving for Internet Gaming | Change from Baseline (T0) Craving for Internet Gaming at 3-month follow-up (T2)
  Craving for Internet Gaming Scale (CIGS) is used to measure respondents' intensity, frequency, duration of their craving, and capability to resist acting on their craving for a particular period of time. It comprises five-item, scoring from 0 to 6 for each item. Respondents with higher scores tend to have higher levels of gaming craving (Cronbach's alpha was .88-.91) (Savci & Griffiths, 2019).
Craving for Internet Gaming | Change from Baseline (T0) Craving for Internet Gaming at 6-month follow-up (T3)
  Craving for Internet Gaming Scale (CIGS) is used to measure respondents' intensity, frequency, duration of their craving, and capability to resist acting on their craving for a particular period of time. It comprises five-item, scoring from 0 to 6 for each item. Respondents with higher scores tend to have higher levels of gaming craving (Cronbach's alpha was .88-.91) (Savci & Griffiths, 2019).
Social support from CSO | Change from Baseline (T0) Social support from CSO at posttest (T1: After intervention)
  The 4-item significant other subscales of the Multidimensional Scale of Perceived Social Support (MSPSS) will be used. It is a self-reporting instrument designed for assessing the level of perceived social support from significant others. The items are scored on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree). The Cantonese version has demonstrated a high internal consistency coefficient with a Cronbach's alpha of .89 (Chou, 2000).
Social support from CSO | Change from Baseline (T0) Social support from CSO at 3-month follow-up (T2)
  The 4-item significant other subscales of the Multidimensional Scale of Perceived Social Support (MSPSS) will be used. It is a self-reporting instrument designed for assessing the level of perceived social support from significant others. The items are scored on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree). The Cantonese version has demonstrated a high internal consistency coefficient with a Cronbach's alpha of .89 (Chou, 2000).
Social support from CSO | Change from Baseline (T0) Social support from CSO at 6-month follow-up (T3)
  The 4-item significant other subscales of the Multidimensional Scale of Perceived Social Support (MSPSS) will be used. It is a self-reporting instrument designed for assessing the level of perceived social support from significant others. The items are scored on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree). The Cantonese version has demonstrated a high internal consistency coefficient with a Cronbach's alpha of .89 (Chou, 2000).
Child-Parent Relationship | Change from Baseline (T0) Child-Parent Relationship at posttest (T1: After intervention)
  The Child-Parent Relationship Scale (C-PRS). The items are scored on a 5-point Likert scale ranging from 1 (very strongly disagree) to 5 (very strongly agree).
Child-Parent Relationship | Change from Baseline (T0) Child-Parent Relationship at 3-month follow-up (T2)
  The Child-Parent Relationship Scale (C-PRS). The items are scored on a 5-point Likert scale ranging from 1 (very strongly disagree) to 5 (very strongly agree).
Child-Parent Relationship | Change from Baseline (T0) Child-Parent Relationship at 6-month follow-up (T3)
  The Child-Parent Relationship Scale (C-PRS). The items are scored on a 5-point Likert scale ranging from 1 (very strongly disagree) to 5 (very strongly agree).
Parental Stress | Change from Baseline (T0) Parental Stress at posttest (T1: After intervention)
  The 17-items Parental Stress Scale (PSS). The items are scored on a 6-point Likert scale ranging from 1 (very strongly disagree) to 6 (very strongly agree).
Parental Stress | Change from Baseline (T0) Parental Stress at 3-month follow-up (T2)
  The 17-items Parental Stress Scale (PSS). The items are scored on a 6-point Likert scale ranging from 1 (very strongly disagree) to 6 (very strongly agree).
Parental Stress | Change from Baseline (T0) Parental Stress at 6-month follow-up (T3)
  The 17-items Parental Stress Scale (PSS). The items are scored on a 6-point Likert scale ranging from 1 (very strongly disagree) to 6 (very strongly agree).
Motivation for treatment | Change from Baseline (T0) Motivation for treatment at posttest (T1: After intervention)
  The 8-item Motivation for Youth's Treatment Scale (MYTS). The items are scored on a 5-point Likert scale ranging from 1 (very strongly disagree) to 5 (very strongly agree).
Motivation for treatment | Change from Baseline (T0) Motivation for treatment at 3-month follow-up (T2)
  The 8-item Motivation for Youth's Treatment Scale (MYTS). The items are scored on a 5-point Likert scale ranging from 1 (very strongly disagree) to 5 (very strongly agree).
Motivation for treatment | Change from Baseline (T0) Motivation for treatment at 6-month follow-up (T3)
  The 8-item Motivation for Youth's Treatment Scale (MYTS). The items are scored on a 5-point Likert scale ranging from 1 (very strongly disagree) to 5 (very strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong College of Technology, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Background] Zhu S, Zhuang Y, Lee P, Li JC, Wong PWC. Leisure and Problem Gaming Behaviors Among Children and Adolescents During School Closures Caused by COVID-19 in Hong Kong: Quantitative Cross-sectional Survey Study. JMIR Serious Games. 2021 May 7;9(2):e26808. doi: 10.2196/26808. PMID 33960954
- [Background] Nielsen P, Christensen M, Henderson C, Liddle HA, Croquette-Krokar M, Favez N, Rigter H. Multidimensional family therapy reduces problematic gaming in adolescents: A randomised controlled trial. J Behav Addict. 2021 Apr 26;10(2):234-243. doi: 10.1556/2006.2021.00022. Print 2021 Jul 15. PMID 33905350
- [Background] Qin L, Cheng L, Hu M, Liu Q, Tong J, Hao W, Luo T, Liao Y. Clarification of the Cut-off Score for Nine-Item Internet Gaming Disorder Scale-Short Form (IGDS9-SF) in a Chinese Context. Front Psychiatry. 2020 May 25;11:470. doi: 10.3389/fpsyt.2020.00470. eCollection 2020. PMID 32528331
- [Background] Siu AMH, Ko FSL, Mak SK. Outcome Evaluation of a Short-Term Hospitalization and Community Support Program for People Who Abuse Ketamine. Front Psychiatry. 2018 Jul 17;9:313. doi: 10.3389/fpsyt.2018.00313. eCollection 2018. PMID 30065669
- [Background] Rustin TA, Tate JC. Measuring the stages of change in cigarette smokers. J Subst Abuse Treat. 1993 Mar-Apr;10(2):209-20. doi: 10.1016/0740-5472(93)90046-5. PMID 8389898
- [Background] Savci, M., & Griffiths, M. D. (2019). The development of the Turkish craving for internet gaming scale (CIGS): A validation study. International Journal of Mental Health and Addiction, 1-18.
- [Background] Chou, K. L. (2000). Assessing Chinese adolescents' social support: The multidimensional scale of perceived social support. Personality and Individual Differences, 28(2), 299-307. https://doi.org/bpjrkw

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05917977/Prot_SAP_000.pdf